CLINICAL TRIAL: NCT01938521
Title: Effects of Red Grape Cells (RGC) Powder on Glycemic and Lipid Control in Patients With Type 2 Diabetes ¬ A Double-blind, Randomized, Placebo Controlled Study
Brief Title: Effects of Red Grape Cells (RGC) Powder in Type 2 Diabetics
Acronym: RGC-T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Prof. Daniela Jakubowicz MD, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0107-13-WOMC
Record Dates: First submitted 2013-09-01; First posted 2013-09-10 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes
Keywords: Red Grape Cells powder (RGC); Placebo (PLA)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Red Grape Cells (RGC) (Experimental): Red Grape Cells (RGC) 1000 mg powder once daily by mouth for three month
  Interventions: Dietary Supplement: Red Grape Cells (RGC)
- Placebo (for Red Grape Cells (RGC)) (Placebo Comparator): Placebo (for Red Grape Cells (RGC)) similar powder to mimic 1000 mg of Red Grape Cells (RGC), once daily by mouth for three month
  Interventions: Dietary Supplement: Placebo (for Red Grape Cells (RGC))

INTERVENTIONS:
Dietary Supplement: Red Grape Cells (RGC) — Red Grape Cells (RGC) 1000 mg powder once daily by mouth for three month
  Other Names: RGC
  Arms: Red Grape Cells (RGC)
Dietary Supplement: Placebo (for Red Grape Cells (RGC)) — Placebo (for Red Grape Cells (RGC)) powder manufactured to mimic Red Grape Cells (RGC) 1000 mg powder
  Other Names: RGC Placebo
  Arms: Placebo (for Red Grape Cells (RGC))

SUMMARY:
The aim of this study is to examine whether the chronic administration during 12 weeks of polyphenols contained in Red Grape Cells (RGC) powder has an effect on mRNA expression of SIRT1 and Clock Genes, on circulating levels of HbA1c, lipids, blood pressure and on postprandial response of glucose, lipids, insulin, C-peptide and GLP-1 in patients with type 2 diabetes .

DETAILED DESCRIPTION:
There is a growing body of evidence demonstrating that polyphenols and specially the most investigated Resveratrol contained in the Red Grape Cells (RGC) exert beneficial effects on several markers of metabolic syndrome i.e. antioxidant, anti-inflammatory, anti-atherosclerotic, vasodilator and antihypertensive activity.

Many of this beneficial metabolic effects of polyphenols, occurs via activation of sirtuin-1 or silent information regulator-1 gene (SIRT1). This gene is expressed in adipose tissue, muscle, endothelium, peripheral blood cells, etc where it plays a pivotal role in the regulation of Circadian Clock Genes (CCG) involved in glucose lipid metabolism, endothelial function, etc .

By activation of SIRT1 and CCG the polyphenols, may influence the circadian secretion of adiponectin, insulin, asymmetric dimethylarginine (ADMA) and other hormones that influence insulin sensitivity, muscular glucose uptake, NO synthesis, nocturnal hepatic glucose production, lipolisis and endothelial function It was shown in several studies in animals and in clinical studies in subjects with metabolic syndrome that SIRT1 expression and its regulation of the CCG, improves insulin sensitivity in skeletal muscle, preventing weight gain; improves pancreatic beta-cell function enhancing insulin secretion and glucose tolerance. It was associated with increased lipolisis in white adipose tissue, decreased glycolysis, increased fatty acid oxidation in skeletal muscle and with increase Nitric Oxide in the endothelium.

Given that polyphenols directly on the clock genes or by enhancing SIRT1 expression appears to counter some of the effects of a high-fat diet, obesity and metabolic syndrome, by protecting against insulin resistance, hyperglycemia, and dyslipidemia and endothelial dysfunction.

It rise the possibility that the polyphenols contained in Red Grape Cells (RGC) by activation SIRT1 may also exert beneficial effects in subjects affected by type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes patients
2. HbA1C > 7 %
3. Duration of diabetes: 0.5 to 20 years
4. Subjects ≥ 30 and ≤70 years of age
5. BMI: 22 to 35 kg/m2
6. Fasting Triglyceride serum level ≥ 150 mg/dl
7. All oral antidiabetic treatments will be allowed, with the exception of thiazolidinediones (glitazones).i.e. pioglitazone (Actos) or rosiglitazone (Avandia). Insulin and no GLP-1 analogs will not be allowed.
8. Normal liver and kidney function
9. Normal thyroid function
10. Acceptable health beside diabetes based on interview, medical history, physical examination, and laboratory tests
11. Willingness to avoid the use of over-the-counter medications, herbs, or supplements throughout the entire study.
12. Willingness to avoid ingestion of any foods containing peanuts, bilberries, blueberries, cranberries, strawberries, raspberries, grapes, grape juice, cocoa powder, dark chocolate, and red wine throughout the entire study
13. Stable physical activity pattern during the three months immediately preceding study
14. Usually wakes up between 06:00 and 07:00 and goes to sleep between 22:00 and 24:00.
15. No shift work within 5 years of the study
16. Did not cross time zones within 1 month of the study
17. Read and understood the informed consent form and signed it voluntarily

    -

Exclusion Criteria:

1. Type 1 diabetes
2. Clinically significant pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, malignant disease
3. Abnormal liver function tests defined as an increase by a factor of at least 2 above the upper normal limit of alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST)
4. Pregnancy or lactation
5. Illicit drug abuse or alcoholism
6. Treatment with thiazolidinediones (glitazones).i.e. pioglitazone (Actos) or rosiglitazone (Avandia).
7. Insulin and or GLP-1 analogs will not be allowed.
8. Anti hyperlipidemic treatment with fibrates. Statins will be allowed
9. Subjects taking anoretic drugs during the month immediately prior to study
10. Subjects on steroid treatment
11. Those with major illnesses, liver, heart, kidney, lung, infectious, neurological, psychiatric, immunological or neoplastic diseases,
12. Those with eating disorders
13. Known hypersensitivity to grapes, soy and/or casein
14. Subjects after bariatric surgery, will be excluded

    -

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Fasting and postprandial Clock Genes expression in peripheral blood cells (PBC) | Fasting and every hour after meal challenge in two occasions : at baseline (day 1) and after 12 weeks of of supplementation with RGC or Placebo .
  In all 40 subjects the effects of 12 weeks supplementation with RGC or placebo will be assessed .The clock gene expression will be measured in peripheral blood cells (PBC), at baseline (Day 1) and again after 12 weeks of supplementation The blood samples will be taken for Clock Genes expression at fasting and after meal challenge every hour until 4 hours

SECONDARY OUTCOMES:
Fasting HbA1c | Fasting blood levels will be taken at baseline and after 12 weeks of supplementation with RGC or placebo
  In all 40 subjects, fasting blood levels for HbA1c, will be measured at baseline and after 12 weeks of supplementation treatment with RGC n=20 or placebo n=20

OTHER OUTCOMES:
fasting and postprandial glucose, Insulin, GLP-1, asymmetric dimethylarginine (ADMA),and lipid plasma levels | The samples will be taken at fasting and every hours until 4 hours after meal challenge, in to occasions at baseline and after 12 week of supplementation with RGC or Placebo
  In all 40 subjects the effects of RGC ingestion or placebo will be evaluated in at baseline and after 12 weeks of supplementation with RGC or placebo. The blood samples will be taken at fasting and every hour up to 4 hours after meal challenge for quantification of Glucose, Insulin, glucagon-like peptide-1 (GLP-1), ADMA and for lipid plasma levels.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Jakubowicz, MD, Principal Investigator — Diabetes Unit E. Wolfson Medical Center. Tel Aviv University
Locations (1):
- Daniela Jakubowicz MD, Holon, Tel Aviv, Israel